CLINICAL TRIAL: NCT02342275
Title: Efficacy and Safety of Propranolol Versus Atenolol on the Proliferative Phase of Infantile Hemangioma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Yi Ji, Doctor, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2014-229
Record Dates: First submitted 2015-01-07; First posted 2015-01-19 (Estimated); Results first posted 2022-06-16 (Actual); Last update posted 2022-06-16 (Actual); Status verified 2022-03

CONDITIONS: Hemangioma
Keywords: Infantile hemangioma; Propranolol; Atenolol; Efficacy; Safety
MeSH Terms: conditions — Hemangioma; Hemangioma, Capillary | interventions — Propranolol; Atenolol

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Propranolol (Active Comparator): Propranolol
  Interventions: Drug: Propranolol
- Atenolol (Active Comparator): Atenolol
  Interventions: Drug: Atenolol

INTERVENTIONS:
Drug: Propranolol — Initiated at a dosage of 1 mg/kg per day divided 3 times daily for 1 week, and then increased to 2 mg/kg per day divided 3 times daily from weeks 2 to 24.
  Other Names: Oral propranolol
  Arms: Propranolol
Drug: Atenolol — Initiated at a dosage of 0.5 mg/kg per day in a single dose for 1 week, and then increased to 1 mg/kg per day in a single dose from weeks 2 to 24.
  Other Names: Oral atenolol
  Arms: Atenolol

SUMMARY:
The purpose of this study is to compare the efficacy of orally administered propranolol versus atenolol in the treatment of potentially disfiguring or functionally threatening IHs.

DETAILED DESCRIPTION:
Currently, propranolol is the preferred treatment for problematic proliferating infantile hemangiomas (IHs). Although propranolol is clearly efficacious, rare side effects, such as hypoglycemia, may be life-threatening. The possibility of propranolol resistance and treatment failure is also important, and highlights the need for employing more established techniques in certain cases.

Nonselective β-adrenergic antagonists, such as propranolol and timolol, are competitive antagonists of catecholamines at the β1- and β2-adrenergic receptors (β-ARs). β2-AR blockade may result in hypoglycemia as a result of decreased glycogenolysis, gluconeogenesis, and lipolysis. Moreover, bronchial hyperreactivity is a direct effect of nonselective β-blockers, resulting in bronchospasms due to pulmonic β2-AR blockade. A solution to minimize many of the side effects of nonselective β-blocker therapy may be the use of more selective β1-blockers such as metoprolol or atenolol, which, at low dosages, have little β2 activity. Unfortunately, there is a paucity of clinical data comparing the efficacy of selective and non-selective β-blocker. Furthermore, because of the broad heterogeneity of IH (e.g., proliferating versus involuting), confounding with other pharmacologic exposures (e.g., corticosteroids), associated complications (e.g., ulceration) and comorbid medical anomalies (e.g., PHACE) that can influence efficiency after IH treatment, observational studies are unable to definitively establish the clinical utility of β-blockers in IH. Thus, questions regarding the efficacy of the subtypes of β-blockers must be answered in randomized controlled trials, which may provide the only way to overcome the selection and ascertainment bias.

The purpose of this study is to compare the efficacy of orally administered propranolol versus atenolol in the treatment of potentially disfiguring or functionally threatening IHs.

ELIGIBILITY:
Inclusion Criteria:

* Patients younger than 24 weeks.
* Presenting a hemangioma with the following characteristics:
* Subcutaneous and/or cutaneous
* Minimum diameter of 1.5 cm on face, 3 cm outside face and 1.5 cm if it is ulcerated.
* Consent of both parents (or the person having parental authority in families)

Exclusion Criteria:

* Infant presenting contraindications for the administration of propranolol or atenolol.
* Hemangioma has been previous treated with corticosteroids, laser, cryotherapy, or only other treatments.
* Patients with an inability to participate or to follow the study treatment and assessment plan.

Max Age: 24 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 377 (Actual)
Dates: Start 2013-10; Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yi Ji, MD, PhD, Principal Investigator — West China Hospital
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ji Y, Chen S, Xu C, Li L, Xiang B. The use of propranolol in the treatment of infantile haemangiomas: an update on potential mechanisms of action. Br J Dermatol. 2015 Jan;172(1):24-32. doi: 10.1111/bjd.13388. Epub 2014 Dec 17. PMID 25196392
- [Background] Ji Y, Chen S, Li K, Li L, Xu C, Xiang B. Signaling pathways in the development of infantile hemangioma. J Hematol Oncol. 2014 Jan 31;7:13. doi: 10.1186/1756-8722-7-13. PMID 24479731
- [Background] Ji Y, Chen S, Li K, Xiao X, Zheng S. Propranolol: a novel antihemangioma agent with multiple potential mechanisms of action. Ann Surg. 2015 Feb;261(2):e52-3. doi: 10.1097/SLA.0000000000000450. No abstract available. PMID 24374526
- [Background] Ji Y, Chen S, Li K, Xiao X, Xu T, Zheng S. Upregulated autocrine vascular endothelial growth factor (VEGF)/VEGF receptor-2 loop prevents apoptosis in haemangioma-derived endothelial cells. Br J Dermatol. 2014 Jan;170(1):78-86. doi: 10.1111/bjd.12592. PMID 24033364
- [Background] de Graaf M, Raphael MF, Breugem CC, Knol MJ, Bruijnzeel-Koomen CA, Kon M, Breur JM, Pasmans SG. Treatment of infantile haemangiomas with atenolol: comparison with a historical propranolol group. J Plast Reconstr Aesthet Surg. 2013 Dec;66(12):1732-40. doi: 10.1016/j.bjps.2013.07.035. Epub 2013 Sep 4. PMID 24011909
- [Background] Raphael MF, de Graaf M, Breugem CC, Pasmans SGMA, Breur JMPJ. Atenolol: a promising alternative to propranolol for the treatment of hemangiomas. J Am Acad Dermatol. 2011 Aug;65(2):420-421. doi: 10.1016/j.jaad.2010.11.056. No abstract available. PMID 21763565
- [Derived] Ji Y, Chen S, Yang K, Zhang X, Zhou J, Li L, Xiang B, Qiu T, Dai S, Jiang X, Lu G, Qiu L, Kong F, Zhang Y. Efficacy and Safety of Propranolol vs Atenolol in Infants With Problematic Infantile Hemangiomas: A Randomized Clinical Trial. JAMA Otolaryngol Head Neck Surg. 2021 Jul 1;147(7):599-607. doi: 10.1001/jamaoto.2021.0454. PMID 33856430

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Propranolol | Atenolol
Started | 190 | 187
Completed | 184 | 182
Not Completed | 6 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Propranolol | Atenolol | Total
Number analyzed (Participants) | 190 | 187 | 377
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 190 | 187 | 377
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: weeks] | 10.2 (4.0) | 9.8 (4.1) | 10.0 (4.047)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 146 | 141 | 287
  Male | 44 | 46 | 90
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  China | 190 | 187 | 377

OUTCOME MEASURES:

1. Primary Outcome: The Primary Outcome Measure Was Any Response at 6 Months
Description: Changes in IH size and color were classified as a complete response, nearly complete response, partial response or no response. The primary outcome measure was any response at 6 months in the intention-to-treat population of all patients who underwent randomization. The any response included compete, nearly complete and partial responses.
  A complete response was defined as no redundant tissue or telangiectasia was identified.
  A nearly complete response was defined as a minimal degree of telangiectasis, erythema and skin thickening.
  A partial response was defined as a size reduction or change in color that did not meet the nearly complete resolution criteria.
Time Frame: 6 month
Measure: Count of Participants; unit: Participants
Arm/Group | Propranolol | Atenolol
Number analyzed (Participants) | 190 | 187
Participants | 178 | 173
Statistical Analysis 1: Comparison: Propranolol vs Atenolol; The sample size required to compare propranolol and atenolol at month 6 was calculated before enrollment. Assuming the ulceration rate in both groups to be 10%, a sample size of180 patients was required for each group to show the noninferiority ofatenolol treatment with a 2-sidedα level of .05 and approximately 90% power; Test type: Non-Inferiority — Assuming that the atenolol on the propranolol response rate does not fall by greater than 15%, the noninferiority margin was selected to be -15%; p < 0.05, Mixed Models Analysis; Odds Ratio (OR) = 0.15 — Treatment Difference=Propranolol vs Atenolol

2. Secondary Outcome: Hemangioma Activity Score (HAS)
Description: HAS was measured at baseline and at 1, 4, 12, and 24 weeks, including the degree of deep swelling, the color of the hemangioma, and the ulceration assessment:
  1. Assessment of the degree of swelling. It was scored as follows:
     * 6 points if the swelling was tense;
     * 4 points if the swelling was'neutral;
     * 2 points when the swelling was reduced by 50% or more at follow-up; or
     * 0 point when there was no more visible swelling at a follow-up.
  2. Assessment of the color of the IH.
     * 5 points if the hemangioma lesion was bright red all over;
     * 3 points if the hemangioma lesion was matte red or reddish-purple;
     * 1 point if the hemangioma lesion was totally or partially gray;
     * 0 points if the hemangioma lesion was totally or partially skin-colored after involution.
  (2) Assessment of the ulceration. -0.5 point for an ulcer ≤1.0 cm2;
  * One point for an ulcer >1.0 cm2 but <25 cm2;
  * Two points for an ulcer ≥25 cm2. The HAS score= (Swelling score + color score)/2 +Ulceration score.
Time Frame: Baseline and at 1, 4, 12, and 24 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Propranolol | Atenolol
Number analyzed (Participants) | 190 | 187
score on a scale
  Baseline | 4.61 (0.82) | 4.54 (0.76)
  Week 1 | 3.31 (0.72) | 3.47 (0.75)
  Week 4 | 2.42 (0.60) | 2.33 (0.65)
  Week 12 | 1.54 (0.79) | 1.54 (0.72)
  Week 24 | 0.82 (0.64) | 0.82 (0.68)

3. Secondary Outcome: Successful Initial Response
Description: A successful initial response was defined as a HAS score decrease at 1 week after treatment.
  A successful initial response was assessed by using HAS in the intention-to-treat population. Previous studies demonstrated that HAS decreases over time after β-blocker treatment, with a dramatic drop occurring in the first week, indicating an immediate therapeutic response. HAS can reflect the rapid effect of β-blocker (either propranolol or atenolol) therapy shortly after initiation.
Time Frame: 1 week after treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Propranolol | Atenolol
Number analyzed (Participants) | 190 | 187
Participants | 171 | 163

4. Secondary Outcome: Complete Ulceration Healing Time
Description: The complete healing time of the ulceration was defined as the time from the first dosage of propranolol or atenolol until complete healing of the hemangioma ulceration (assessed up to 6 months). Ulceration is defined as a break in the integrity of the hemangioma surface epithelium (or skin) with or without infection. The information included the extent of ulceration, complications of ulceration, prior duration of ulceration (before treatment), concurrent treatments, and complete healing time. Prior duration of ulceration was defined as the time from the first sign of ulceration until before β-blocker treatment. The complete healing time of the ulceration was defined as the time from the first dosage of propranolol or atenolol until complete healing of the hemangioma ulceration. Concurrent treatments, including oral pain medication, oral antibiotics, topical ointment antibiotics and/or wound dressings, were permitted to treat ulcerated IH and were recorded.
Time Frame: from the first dosage of propranolol or atenolol until complete healing ofthe hemangioma ulceration.
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Propranolol | Atenolol
Number analyzed (Participants) | 190 | 187
weeks | 4.94 (2.16) | 4.82 (1.75)

5. Secondary Outcome: Rebound Rate
Description: Regrowth of more than 20% in hemangioma appearance (including changes in color and/or volume) after stopping the medication was considered significant rebound. The inclusion criteria for rebound analysis were as follows: (1) patients who completed 6 months of treatment and (2) patients who discontinued therapy or were tapering treatment after achieving an any response. The exclusion criteria were as follows: (1) patients who were noncompliant with treatment and (2) patients who did not respond to treatment. Whether a patient had hemangioma rebound was based on the site investigators' assessments after the week 24 treatment. In patients with significant rebound, reinitiation of systemic therapy (either propranolol or atenolol) was recommended. Minor rebound, which was defined as those patients in whose rebound was noted but no reinitiation of systemic therapy or further treatment was necessary, was not included in the analysis.
Time Frame: between weeks 24 and 96
Population: Data only included patients who attempted to discontinue β-blockers according to the treatment plan between weeks 24 and 96
Measure: Count of Participants; unit: Participants
Arm/Group | Propranolol | Atenolol
Number analyzed (Participants) | 170 | 160
Participants | 19 | 12

6. Secondary Outcome: Number of Participants With Complete/Nearly Complete Response (96 Week)
Description: A complete/nearly complete response at week 96 was considered median-term efficacy.
Time Frame: 96 week
Measure: Count of Participants; unit: Participants
Arm/Group | Propranolol | Atenolol
Number analyzed (Participants) | 190 | 187
Participants | 156 | 149

ADVERSE EVENTS:
Time Frame: Adverse events during the initial 6 months of treatment were compared between the 2 groups.
Arm/Group | Propranolol | Atenolol
All-Cause Mortality (participants affected / at risk) | 0/190 | 0/187
Serious Adverse Events (participants affected / at risk) | 5/190 | 3/187
Other Adverse Events (participants affected / at risk) | 128/190 | 80/187
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Propranolol (N=190) | Atenolol (N=187)
Sleep disturbance (Nervous system disorders) | 2 | 0 — Severe sleep disturbance was defined as sleep disturbance that did not disappear or was not relieved after treatment administration was altered (eg, earlier evening dose or a decrease in daily dose)
Bronchiolitis (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 1
Viral upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Propranolol (N=190) | Atenolol (N=187)
Diarrhea (Gastrointestinal disorders) | 25 | 27
Sleep disturbance (Nervous system disorders) | 25 | 9
Agitation (Psychiatric disorders) | 16 | 5
Cool extremities (Blood and lymphatic system disorders) | 14 | 6
Bradycardia (Cardiac disorders) | 13 | 9
Vomiting (Gastrointestinal disorders) | 7 | 5
Hypotension (Vascular disorders) | 9 | 4
Bronchiolitis (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Decreased appetite (Gastrointestinal disorders) | 7 | 5
Constipation (Gastrointestinal disorders) | 4 | 6
Viral upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-01): https://cdn.clinicaltrials.gov/large-docs/75/NCT02342275/Prot_SAP_000.pdf